CLINICAL TRIAL: NCT02452060
Title: Randomized, Double-blind, Placebo Controlled Study on the Effect of a Single Postoperative Administration of Low Dose Ketamine After Gastric Bypass and Gastrectomy Surgeries
Brief Title: Study on the Use of Low Dose Ketamine After Gastric Bypass and Gastrectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14-00472
Record Dates: First submitted 2015-04-16; First posted 2015-05-22 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Pain; Postoperative Depression
Keywords: perioperative period; pain; gastric bypass
MeSH Terms: conditions — Pain | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment/placebo (Placebo Comparator): saline infusion
  Interventions: Other: Placebo Comparator
- treatment (Experimental): ketamine (0.4mg/kg)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — 0.4mg/kg infusion
  Other Names: ketalar
  Arms: treatment
Other: Placebo Comparator — 0.4mg/kg infusion
  Other Names: Saline Infusion
  Arms: treatment/placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, two-arm parallel, single-center study. One hundred subjects (50 in each arm) will be enrolled. Subjects, between the ages 18 and 65, undergoing laparoscopic gastric bypass or sleeve gastrectomy will be recruited and consented during the preadmission visit prior to surgery.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, two-arm parallel, single-center study. One hundred subjects (50 in each arm) will be enrolled. Subjects, between the ages 18 and 65, undergoing laparoscopic gastric bypass or sleeve gastrectomy will be recruited and consented during the preadmission visit prior to surgery. Eligible subjects will be randomized to one of the two treatment group in a 1:1 ratio to receive either IV ketamine (0.4mg/kg) or matching placebo. Both men and women will be recruited, and there is no limitation as to racial and ethnic origin. In the PACU, patients will receive either 0.4mg/kg IV ketamine or placebo. All patients will also receive standard post-anesthetic monitoring and care, as well as routine care after transfer out of the PACU. Patients are followed until the date of discharge, and endpoints (see below) are collected from patient reports as well as from medical charts. During their hospital stay (and once after their discharge from the hospital), patients will fill out five questionnaires which provide estimates of their postoperative pain control, mood and function, and quality of postsurgical recovery. An additional component of the study, which is entirely optional, is to obtain patient serum samples (about two teaspoons) in the operating room and 15 minutes and 4 hours after ketamine infusion. The investigators will use these samples to assess levels of IL-1, IL-6, TNF-α, and BDNF, which are markers for pain. In addition, with patient consent, the investigators will also store serum samples for future research use to measure other cytokines and neurotrophic factors and molecular markers associated with pain and depression.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, >18 years, <65 years, who will undergo gastric bypass or sleeve gastrectomy.
2. Subject is non-lactating and is either:

   * Not of childbearing potential; or
   * Of childbearing potential but is not pregnant at time of baseline as determined by pre-operative pregnancy testing.
3. Subject is ASA physical status 1, 2, or 3.
4. Subject who is deemed medically stable

Exclusion Criteria:

1. <18 years of age; >65 years of age
2. Pregnant or breastfeeding
3. Does not speak or understand English (the study forms used are copy-righted in English)
4. Cognitively impairment (by history) or clinical signs of altered mental status
5. History of misuse or abuse of ketamine
6. History of chest pain or chest pain in the PACU
7. Use of a medication that interferes with metabolism of ketamine within the last 24 hours
8. A diagnosis of schizophrenia and/ or a history of chronic antipsychotic medication use
9. History of head trauma
10. History of intracranial mass or hemorrhage
11. History of stroke
12. History of cardiac arrhythmia
13. Subject for whom ketamine is contraindicated
14. Unwillingness to give informed consent according to HIC guidelines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-04-13 (Actual); Study Completion 2017-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jing Wang, MD, PHD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Wang J, Echevarria GC, Doan L, Ekasumara N, Calvino S, Chae F, Martinez E, Robinson E, Cuff G, Franco L, Muntyan I, Kurian M, Schwack BF, Bedrosian AS, Fielding GA, Ren-Fielding CJ. Effects of a single subanaesthetic dose of ketamine on pain and mood after laparoscopic bariatric surgery: A randomised double-blind placebo controlled study. Eur J Anaesthesiol. 2019 Jan;36(1):16-24. doi: 10.1097/EJA.0000000000000860. PMID 30095550

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment/Placebo | Treatment
Started | 46 | 44
Completed | 46 | 44
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo Comparator: 0.4mg/kg saline infusion
- Total: Total of all reporting groups
Arm/Group | Placebo | Ketamine | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 44 | 90
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 33 | 62
  Male | 17 | 11 | 28
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 8 | 9 | 17
  White | 37 | 35 | 72
  Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scores
Description: VAS Scores will be assessed on Day of Surgery (DOS), Post-op Day (POD) 1, 2 and 7. If patients have been discharged, coordinators will contact patient by home.
Time Frame: Baseline (DOS) to 7 days (Post Op)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment/Placebo | Treatment
Number analyzed (Participants) | 46 | 44
score on a scale | 1.45 (.23) | 1 (0.18)

2. Secondary Outcome: Length of Stay During Hospitalization
Description: LOS will be recorded from medical record.
Time Frame: 8 days
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Treatment/Placebo | Treatment
Number analyzed (Participants) | 46 | 44
Days | 1.3 [1 to 2] | 1.2 [1 to 1.9]

3. Other Pre Specified Outcome: Opioid Usage Per Hour During the PACU Stay Before and After Ketamine Infusion
Description: Length of stay and opioid usage will be recorded from electronic medical chart
Time Frame: 8 Days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Opioid Usage Per Day Throughout the Hospital Stay
Description: recorded from medical chart
Time Frame: 8 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Time to Out of Bed to Chair (OOB)
Description: Patient will be asked to record and report the time to OOB
Time Frame: 7 Days
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Spirometry Use 4 Hours After the Termination of Ketamine Infusion
Description: Spirometry use will be assessed by a study team member to determine whether the patient is meeting the goal set by the surgical team 4 hours after ketamine infusion.
Time Frame: 1 day
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Change in Serum Level of IL-1 After Ketamine Infusion
Description: changes in serum levels of IL-1, which will be collected at baseline (in the OR preoperatively), and 15 min and 4 hours after the termination of ketamine infusion.
Time Frame: 1 day
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Survey Scores - McGill's Short Form
Description: Change in survey scores -- McGill's short form
Time Frame: Pre-op,Day of Surgery through Post-op Day 8
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Survey Scores - Becks Depression Index (BDI)
Description: Change in survey scores for Becks Depression Index (BDI)
Time Frame: Pre-op,Day of Surgery through Post-op Day 8
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Survey Scores - QoR15
Description: Change in scores for Quality of Recovery 15 - QoR15
Time Frame: Pre-op,Day of Surgery through Post-op Day 8
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Survey Scores - MADRS
Description: Change in scores for MADRS
Time Frame: Pre-op,Day of Surgery through Post-op Day 8
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Change in Serum Level of IL-6 After Ketamine Infusion
Description: as for outcome 7
Time Frame: 1 day
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Change in Serum Level of TNF-α After Ketamine Infusion
Description: as for outcome 7
Time Frame: 1 day
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Change in Serum Level of BDNF After Ketamine Infusion
Description: as for outcome 7
Time Frame: 1 day
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 Year
Description: 0
Arm/Group | Treatment/Placebo | Treatment
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 9/46 | 7/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment/Placebo (N=46) | Treatment (N=44)
dizziness/lightheadedness (General disorders) | 1 (1) | 5 (5)
nausea (General disorders) | 2 (2) | 2 (2)
euphoria (General disorders) | 2 (2) | 0 (0)
visual hallucination (Psychiatric disorders) | 2 (2) | 0 (0)
headache (General disorders) | 1 (1) | 0 (0)
Dysphoria (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT02452060/Prot_SAP_000.pdf